CLINICAL TRIAL: NCT00425932
Title: Impact of Rituximab on Magnetic Resonance Imaging Evidence of Synovitis and Bone Lesions in Patients With Moderate or Severe Rheumatoid Arthritis
Brief Title: Impact of Rituximab on MRI Evidence of Disease Activity in Patients With Moderate to Severe Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gaylis, Norman B., M.D. (Individual)
Collaborators: Oklahoma Medical Research Foundation (Other); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: U3900s
Record Dates: First submitted 2007-01-22; First posted 2007-01-24 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Magnetic Resonance Imaging; Rituximab; Low Field MRI; Biomarkers
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Rituximab/Placebo (No Intervention): Patients will be randomized at Baseline to either Placebo or Rituximab. At Week 24 and up to Week 48 if patient DAS28 score is >2.6, patient will be retreated with open label Rituximab.
- Open Label (Active Comparator): At Week 24 or any time up to Week 48 if the Patient DAS 28 > 2.6 patients will be retreated with 1000 mg IV at Day and Day 15.
  Interventions: Biological: Rituximab

INTERVENTIONS:
Biological: Rituximab — At Week 24 or any time up to Week 48 if the Patient DAS 28 > 2.6 patients will be retreated with 1000 mg IV at Day and Day 15.
  Other Names: Rituxan
  Arms: Open Label

SUMMARY:
The purpose of this study is to further investigate rituximab in the treatment of rheumatoid arthritis and to evaluate magnetic resonance imaging of the joints as a possible method to improve the evaluation of treatments.

DETAILED DESCRIPTION:
Rituximab is a monoclonal antibody that has been approved for the treatment of non-Hodgkin's B cell lymphoma (a type of cancer) and for certain patients with rheumatoid arthritis (RA) by the Food and Drug Administration (FDA). To date, more than 1000 subjects with rheumatoid arthritis have received rituximab in clinical studies.

Magnetic resonance imaging (MRI) is a modern and sensitive method of looking at joints in people with rheumatoid arthritis. It uses a magnetic field to create an image. The MRI takes an image in 3 dimensions and this provides a better picture for a physician to see more details.

There are two treatment groups in this study with equal numbers of patients assigned to each group. All the patients will receive their baseline Methotrexate and two intravenous infusions 2 weeks apart of one of the following:

* 1000 mg rituximab or
* placebo. Patients outcomes will be compared between the 2 groups. After week 24 (open label phase), the patients will receive rituximab if rheumatoid arthritis remains active.

All the patients will have MRI of their dominant hand and wrist with and without gadolinium performed at baseline, 12, 24 and 48 weeks on 1.5 Tesla MRI . Some patients will also have additional MRI of the same hand and wrist without gadolinium at the same time points on 0.2 Tesla MRI. Comparison of the images from the two machines will be performed.

Various blood biomarkers will also be examined, compared between the 2 treatment groups and correlated with the MRI results.

ELIGIBILITY:
Inclusion Criteria

* Able and willing to give written informed consent
* Age 18-80 years
* Must have active rheumatoid arthritis for at least 12 weeks, but no more than 5 years.
* Must be receiving treatment on an outpatient basis
* Must have > 8 tender and swollen joints
* Must have negative serum pregnancy test
* Must have an inadequate response to MTX
* Must have elevated serology parameters
* Must have Positive RF or anti-CCP antibody, or radiographic evidence of at least one joint with definite erosion attributable to RA.
* Stable use of Corticosteroids is permitted
* Stable use of NSAIDs is permitted

Exclusion Criteria:

* History of or current inflammatory joint disease
* Functional class IV
* Any surgical procedure within 12 weeks
* Lack of peripheral venous access.
* Pregnancy or breast feeding.
* Significant cardiac or pulmonary disease.
* Evidence of significant uncontrolled concomitant disease
* Positive HIV
* Known active infection of any kind
* History of deep space/tissue infection
* History of recurrent significant infection
* Concomitant malignancies or previous malignancies
* Any neurological, vascular or systemic disorder
* History of drug, alcohol, or chemical abuse
* Inability to comply with study and follow-up procedures
* History of a severe allergic or anaphylactic reaction to a biologic agent
* Previous treatment with more than one biologic agent for RA. Patients must not have received a biologic agent within 2 months prior to the Baseline visit, except for etanercept, abatacept and anakinra for which a one month washout prior to Baseline visit is acceptable
* Previous treatment with an anti-alpha 4 integrin antibody or co-stimulation modulator.
* Previous treatment with any cell depleting therapies.
* Treatment with any investigational agent within 28 days
* Receipt of a live/attenuated vaccine within 28 days
* Ongoing use of high dose steroids (>10mg/day)
* Inra-articular or parental glucocorticoids within 4 weeks prior to baseline.
* Intolerance or contraindications to i.v. glucocorticoids.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-02; Primary Completion 2011-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
The primary endpoint fo the trial is change in 1.5 Tesla MRI erosion score (RAMRIS system) from baseline to Week 24. | 24 weeks

SECONDARY OUTCOMES:
Change from Baseline in 1.5 Tesla MRI synovitis score (RAMRIS system) at Week 12. | 12 weeks
Change from Baseline in 1.5 Tesla MRI bone edema and total score (RAMRIS system) at Week 24. | 24 weeks
Change from Baseline in 1.5 Tesla MRI bone edema, bone erosion and total score (RAMRIS system) at Week 12 and Week 48. | 12 and 48 weeks
Proportion of patients at Week 48 without new bone erosions on 1.5 Tesla MRI. | 48 weeks
Change from baseline in total Genant modified Sharp score on conventional radiographs at Week 24 and 48. | 24 and 48 weeks
Change in Disease Activity Score (DAS 28) from Baseline to Week 24 and 48. | 24 and 48 weeks
ACR remission and responder rates (20%, 50%, &)%) at Week 24 and 48. | 24 and 48 weeks
Change from Baseline in functional assessments according to the HAQ scores at 24 and 48 Weeks. | 24 and 48 weeks
Difference between relative results from conventional high-field strength 1.5 Tesla MRI and 0.2 Tesla dedicated extremity MRI in detection and grading of bone erosions, bone edema, and synovitis at Baseline and in Week 12,24, and 48 (C-scan validation). | 12, 24 and 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Norman B Gaylis, MD, Principal Investigator — Arthritis & Rheumatic Disease Specialties; Ewa Olech, M.D., Principal Investigator — Oklahoma Medical Research Foundation
Locations (6):
- United States (6):
  - Guillermo Valenzuela MD, Fort Lauderdale, Florida
  - Drs. Charles Kahn and Wayne Riskin, Hollywood, Florida
  - Arhtritis & Rheumatic Disease Specialties, Miami, Florida
  - Arthritis and Rheumatology Clinics of Kansas, Wichita, Kansas
  - McBride Clinic Orthopedic Center, Oklahoma City, Oklahoma
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma

REFERENCES:
- [Derived] Peterfy CG, Olech E, DiCarlo JC, Merrill JT, Countryman PJ, Gaylis NB. Monitoring cartilage loss in the hands and wrists in rheumatoid arthritis with magnetic resonance imaging in a multi-center clinical trial: IMPRESS (NCT00425932). Arthritis Res Ther. 2013 Mar 20;15(2):R44. doi: 10.1186/ar4202. PMID 23514433